CLINICAL TRIAL: NCT02413710
Title: A Randomized, Controlled, Parallel Study to Assess the Effects of Soy Protein on Body Composition and General Health Parameters in Healthy Children
Brief Title: Effects of Soy Protein on Body Composition and General Health in Healthy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DuPont Nutrition and Health (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BIO-1501
Record Dates: First submitted 2015-03-17; First posted 2015-04-10 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Generally Healthy Kids Consumption Soy Protein Foods as Part of Daily Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Protein Group (Active Comparator): Subjects will be instructed on the 2010 Dietary Guidelines for Americans including publically available information from the United States Department of Agricultural (USDA) MyPlate program (www.choosemyplate.gov). Subjects in this intervention group will not receive study provided foods.
  Interventions: Behavioral: Dietary Guidance
- Soy Protein Group (Experimental): Subjects will be instructed on the 2010 Dietary Guidelines for Americans including publically available information from the USDA MyPlate program (www.choosemyplate.gov) with the incorporation of two servings of study food providing soy protein per day.
  Interventions: Other: Soy protein containing foods

INTERVENTIONS:
Other: Soy protein containing foods — Daily consumption of 2 food products, each providing 15g of soy protein per day.
  Arms: Soy Protein Group
Behavioral: Dietary Guidance — Subjects will be instructed on the 2010 Dietary Guidelines for Americans including publically available information from the United States Department of Agricultural (USDA) MyPlate program (www.choosemyplate.gov). Subjects in this intervention group will not receive study provided foods.
  Arms: Usual Protein Group

SUMMARY:
The aim of this clinical trial is to assess the effects of daily consumption of soy protein foods on body composition, general health status and dietary intake outcomes in generally healthy children.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, 8-11 years of age, inclusive.
2. Subject is judged to be in good health on the basis of medical history.
3. Subject is a regular consumer (5 out of 7 d) of breakfast and snacks.
4. Subject has a BMI-for-age within the 75th and 95th percentile (Appendix 3).
5. Subject is willing to follow dietary changes consistent with the Dietary Guidelines for Americans 2010 throughout the study period (Appendix 5).
6. Subject/guardian understands the study procedures and signs forms providing assent/informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigators.

Exclusion Criteria:

1. Subject has a diagnosis of attention deficit disorder, with or without hyperactivity.
2. Subject requires special educational services related to cognitive or attentional disorders, neurologic diseases, and physical disabilities.
3. Subject is a girl who has begun menses.
4. Subject is at Tanner Stage IV or higher, as described by parent/guardian per self-assessment questionnaire (Appendix 2).
5. Subject has a history or presence of a clinically relevant cardiac, renal, hepatic, endocrine (including diabetes mellitus), pulmonary, biliary, gastrointestinal, pancreatic, or neurologic disorder.
6. Subject has a known allergy or sensitivity to the study foods.
7. Use of sleep aids within 2 weeks of visit 1 (week -1) and throughout the study.
8. Subject has extreme dietary habits, in the judgment of the Investigator.
9. Subject has used any weight loss supplements, programs, or meal replacement products (within 2 weeks of visit 1, week -1) intended to alter body weight (Appendix 1).
10. Subject has a history of an eating disorder (e.g., anorexia nervosa, bulimia nervosa or binge eating) diagnosed by a health professional.
11. Involvement in any clinical trial within 30 d prior to the screening visit.
12. Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
change in body composition | week 0, week 12
  DXA

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis Clinical Research, Addison, Illinois, United States